CLINICAL TRIAL: NCT07280689
Title: Mejorar la empatía Hacia el Mayor Mediante la simulación de la Vejez
Brief Title: Effects of an Aging Simulation Suit on Clinical Empathy in Healthcare Professionals Working in Long-Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Participating Nursing Homes in Madrid and Asturias, Spain (Unknown)
Responsible Party: Principal Investigator, Sergio Serrada Tejeda, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2711201916919
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Aging; Empathy Skills
Keywords: Clinical empathy; GERT suit; randomized controlled trial; Healthcare professionals; Aging simulation suit

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: a control group that received a theoretical educational session on aging and empathy, and an experimental group that received the same session plus an immersive experience using an aging simulation suit.
Masking Description: Due to the nature of the educational intervention, neither participants nor investigators were blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Aging Simulation Suit + Educational Session (Experimental): Participants received a theoretical session on aging, functional limitations, and empathy in healthcare, followed by an immersive experience using the GERT aging simulation suit. The suit replicates the physical and sensory limitations of aging, allowing participants to perform everyday tasks while experiencing the challenges faced by older adults.
  Interventions: Behavioral: Experimental: Aging Simulation Suit + Educational Session; Behavioral: Control: Educational Session Only
- Control: Educational Session Only (Active Comparator): Participants received the same theoretical session on aging, functional limitations, and empathy in healthcare as the experimental group, but did not use the aging simulation suit.
  Interventions: Behavioral: Control: Educational Session Only

INTERVENTIONS:
Behavioral: Experimental: Aging Simulation Suit + Educational Session — Immersive training session using the GERT aging simulation suit (Niederstotzingen, Germany), designed to reproduce age-related physical and sensory limitations. Participants performed common daily activities (e.g., walking, climbing stairs, dressing, interacting with others) while wearing the suit to experience the physical challenges of aging. This activity was followed by a short debriefing and group reflection aimed at enhancing empathy and awareness toward older adults.
  Arms: Experimental: Aging Simulation Suit + Educational Session
Behavioral: Control: Educational Session Only — A structured theoretical session covering topics such as aging processes, functional limitations, and the importance of empathy in healthcare and long-term care contexts. Delivered to all participants in both study arms, serving as the baseline educational component for the control and experimental groups.

SUMMARY:
This randomized controlled trial examined the effects of using an aging simulation suit on empathy levels among healthcare professionals working in long-term care facilities. A total of 82 participants from four nursing homes in Madrid and Asturias were randomly assigned to an experimental group or a control group. The experimental group received a theoretical session on aging and empathy, followed by an immersive experience using the GERT aging simulation suit, which replicates age-related physical and sensory limitations. The control group attended only the theoretical session.

Empathy was assessed before and after the intervention using the Interpersonal Reactivity Index (IRI) and the Jefferson Scale of Empathy - Health Professions version (JSPE-HPS). Results showed significant improvements in the JSPE-HPS total score and in its Perspective Taking and Compassionate Care dimensions in the experimental group, indicating that the immersive experience enhanced both cognitive and affective components of clinical empathy. No significant changes were observed in the IRI scores.

These findings suggest that experiential learning through aging simulation can effectively strengthen empathy in active healthcare professionals, promoting more person-centered and compassionate care for older adults in long-term care settings.

DETAILED DESCRIPTION:
Aging is accompanied by physiological, structural, and psychosocial changes that affect mobility, sensory functions, and interaction with the environment. Healthcare professionals working in long-term care facilities play a crucial role in supporting the physical, emotional, and social well-being of older adults. Empathy, understood as the ability to understand and share another person's feelings, is a key component of effective therapeutic relationships and person-centered care.

Traditional empathy training for healthcare providers often relies on lectures, role-playing, or observation of patient interactions. However, there is limited evidence regarding the impact of immersive simulation-based methods on empathy among active healthcare professionals. The use of aging simulation suits, which reproduce the physical and sensory limitations of older adults, has emerged as an innovative educational tool to promote understanding of the aging experience and improve empathic attitudes toward older persons.

This randomized controlled trial was designed to evaluate the effect of an aging simulation suit (GERT, Niederstotzingen, Germany) on levels of clinical empathy among healthcare professionals working in long-term care facilities. Participants were randomly assigned to one of two groups:

Experimental Group: Received a theoretical educational session on aging, functional limitations, and the role of empathy in care, followed by a practical session using the aging simulation suit. During the simulation, participants performed daily living tasks (e.g., walking, climbing stairs, dressing, interacting with others) while experiencing the physical restrictions associated with advanced age.

Control Group: Received only the theoretical session on aging and empathy without the immersive simulation experience.

Empathy was assessed pre- and post-intervention using two validated instruments:

Interpersonal Reactivity Index (IRI) - measures cognitive and emotional dimensions of general empathy.

Jefferson Scale of Empathy - Health Professions version (JSPE-HPS) - evaluates empathy specifically in clinical contexts.

Data analysis was conducted using repeated-measures ANOVA to assess within- and between-group differences over time.

Main findings: The experimental group showed significant increases in total JSPE-HPS scores and in the subscales Perspective Taking and Compassionate Care, whereas the control group showed no significant changes. No significant differences were observed in IRI scores. These results indicate that immersive experiential learning through the use of an aging simulation suit can enhance both cognitive and affective aspects of empathy in healthcare professionals.

The study was approved by the Ethics Committee of Universidad Rey Juan Carlos and conducted in accordance with the Declaration of Helsinki and ICH Good Clinical Practice guidelines.

This research supports the integration of simulation-based empathy training in continuing professional education for healthcare workers in long-term care, promoting more compassionate, person-centered care for the aging population.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professional (nurse, nursing assistant, occupational therapist, physiotherapist, physician, psychologist, or social worker).
* Currently working in a long-term care or nursing home facility with direct contact with residents.
* Willing to participate voluntarily during working hours.
* Signed written informed consent.

Exclusion Criteria:

* Failure to provide written informed consent.
* No direct patient contact with older adults.
* Any physical or cognitive limitation that would prevent safe participation in the aging simulation experience.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in total score on the Jefferson Scale of Empathy - Health Professions version (JSPE-HPS) | Pre-intervention (baseline) and immediately post-intervention (same day)
  Mean difference in total Jefferson Scale of Physician Empathy - Health Professional Student version (JSPE-HPS) score between baseline (pre-intervention) and post-intervention for each study group. The JSPE-HPS measures clinical empathy in healthcare professionals and consists of 20 items, with total scores ranging from 20 to 140; higher scores indicate higher empathy (better outcome). The primary analysis was performed using repeated-measures ANOVA to examine time effects and the group × time interaction.

SECONDARY OUTCOMES:
Change in Perspective Taking subscale of the JSPE-HPS | Pre-intervention and immediately post-intervention (same day)
  Mean pre/post difference in the Perspective Taking subscale of the Jefferson Scale of Physician Empathy - Health Professional Student version (JSPE-HPS). The JSPE-HPS consists of 20 items rated on a 7-point Likert scale (total score range 20-140). The Perspective Taking subscale comprises 10 items, with subscale scores ranging from 10 to 70. This subscale assesses cognitive empathy, and higher scores indicate higher levels of empathy (better outcome). Differences were analyzed using repeated-measures ANOVA, including the group × time interaction.
Change in Compassionate Care subscale of the JSPE-HPS | Pre-intervention and immediately post-intervention (same day)
  Mean pre/post difference in the Compassionate Care subscale of the Jefferson Scale of Physician Empathy - Health Professional Student version (JSPE-HPS). This subscale assesses affective aspects of clinical empathy, with higher scores indicating higher empathy (better outcome). Differences were analyzed using repeated-measures ANOVA, including the group × time interaction.
Change in Standing in the Patient's Shoes subscale of the JSPE-HPS | Pre-intervention and immediately post-intervention (same day)
  Mean pre/post difference in the Standing in the Patient's Shoes subscale of the Jefferson Scale of Physician Empathy - Health Professional Student version (JSPE-HPS). This subscale assesses the ability to adopt the patient's perspective, with higher scores indicating higher empathy (better outcome). Differences were analyzed using repeated-measures ANOVA, including the group × time interaction.
Change in total score on the Interpersonal Reactivity Index (IRI) | Pre-intervention and immediately post-intervention (same day)
  Mean difference in total Interpersonal Reactivity Index (IRI) score between pre- and post-intervention. The IRI is a 28-item measure distributed across four subscales (Perspective Taking, Fantasy, Empathic Concern, and Personal Distress), with total scores ranging from 0 to 112. Higher total scores indicate greater empathic disposition. Data were analyzed using repeated-measures ANOVA to evaluate time effects and the group × time interaction.
Change in IRI subscale scores (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) | Pre-intervention and immediately post-intervention (same day)
  Mean pre/post difference in each of the four Interpersonal Reactivity Index (IRI) subscales (Perspective Taking, Fantasy, Empathic Concern, and Personal Distress), each consisting of 7 items with scores ranging from 0 to 28. For Perspective Taking, Fantasy, and Empathic Concern, higher scores indicate greater empathy (better outcome), whereas for Personal Distress, higher scores indicate greater self-oriented distress (worse outcome). Each subscale was analyzed separately using repeated-measures ANOVA to examine time effects and the group × time interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa María Martínez Piédrola, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset includes information from a small group of healthcare professionals that could potentially allow identification of participants. Only aggregated and anonymized summary results will be published in scientific journals and conference presentations.

REFERENCES:
- [Result] Lee K, Han A, Kim TH. Effectiveness of Simulation-Based Empathy Enhancement Program for Caregivers (SEE-C) Evaluated by Older Adults Receiving Care. Int J Environ Res Public Health. 2021 Jul 23;18(15):7802. doi: 10.3390/ijerph18157802. PMID 34360095
- [Result] Pira GL, Ruini C, Vescovelli F, Banos R, Ventura S. Could Empathy Be Taught? The Role of Advanced Technologies to Foster Empathy in Medical Students and Healthcare Professionals: A Systematic Review. J Med Syst. 2025 Jan 14;49(1):6. doi: 10.1007/s10916-025-02144-9. PMID 39806022
- [Result] Ebm C, Sarti R, Panico P, Pagliotta M, Vinci V, Oldani S. Enhancing compassion in medical education - a comparative study of the efficacy of clinical clerkships versus simulation-based training methodologies. BMC Med Educ. 2025 Feb 4;25(1):181. doi: 10.1186/s12909-025-06687-w. PMID 39905468
- [Result] Halton C, Cartwright T. Walking in a Patient's Shoes: An Evaluation Study of Immersive Learning Using a Digital Training Intervention. Front Psychol. 2018 Nov 12;9:2124. doi: 10.3389/fpsyg.2018.02124. eCollection 2018. PMID 30483174